CLINICAL TRIAL: NCT01229527
Title: Comparison Between Two Different Dosages of Remifentanil Administered by PCSA (Patient Controlled Sedation and Analgesia) and Meperidine During Colonoscopy: A Randomized Double-Blind Trial
Brief Title: Comparison Between Two Different Dosages of Remifentanil During Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Agostoni Massimo, Medical Doctor, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PCSA/Remi 2009
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Remifentanil; Sedation
MeSH Terms: interventions — Remifentanil; Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Remifentanil RS1 (Experimental)
  Interventions: Drug: Remifentanil
- Remifentanil RS2 (Experimental)
  Interventions: Drug: Remifentanil
- Meperidine (Active Comparator)
  Interventions: Drug: Meperidine

INTERVENTIONS:
Drug: Remifentanil — Patient receive a bolus of Remifentanil (0,5 mcg/Kg) before the procedure and the PCSA pump is set to inject further bolus doses of 0,5 mcg/Kg every time the patient presses its button.
  Arms: Remifentanil RS1
Drug: Remifentanil — Patient receive a bolus of Remifentanil (0,8 mcg/Kg) before the procedure and the PCSA pump is set to inject further bolus doses of 0,8 mcg/Kg every time the patient presses its button.
  Arms: Remifentanil RS2
Drug: Meperidine — Patient receive a bolus of Meperidine (0,7 mg/Kg) before the procedure and the PCSA pump with saline (sham PCSA) is connected.
  Arms: Meperidine

SUMMARY:
The purpose of this randomized double-blind trial is to define the correct dosage of Remifentanil during operative and diagnostic endoscopic procedures. In particular we want to analyze if the administration of Remifentanil by PCSA (Patient Controlled Sedation and Analgesia) is a good method during colonoscopy, evaluating pain control, discharge time and side effects.

90 patients undergoing colonoscopy will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* Diagnostic and Operative Colonoscopy
* ASA Physical Status I-II

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil RS1 | Remifentanil RS2 | Meperidine
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil RS1 | Remifentanil RS2 | Meperidine | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 19 | 62
  >=65 years | 10 | 7 | 11 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 58.93 (11.15) | 55.10 (11.82) | 60.37 (10.48) | 58.13 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 16 | 40
  Male | 17 | 19 | 14 | 50
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Discharge Time, the Time to Reach a Modified Aldrete Score ≥18
Description: Ten key parameters (Activity, Respiration, Circulation, Consciousness, O2 Saturation, Dressing, Pain, Ambulation, Fasting-feeding, Urine Output)are included in the Modified Aldrete Score. The maximum and minimum score for each parameter is respectively 2 and 0. The maximum total score is 20 and patient can be discharged when the total score is ≥18.
Time Frame: > 0 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remifentanil RS1 | Remifentanil RS2 | Meperidine
Number analyzed (Participants) | 30 | 30 | 30
minutes | 0 [0 to 1] | 0 [0 to 1] | 2 [1 to 4]

2. Secondary Outcome: Patient's Satisfaction
Description: The degree of satisfaction about the quality of sedation was measured with VAS (Visual Analog Scale) where 0 means no satisfaction and 100 means maximum satisfaction.
Time Frame: After the end of colonoscopy (when patients were completely awake) and 24 h after the procedure via telephone
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remifentanil RS1 | Remifentanil RS2 | Meperidine
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | 95.87 (9.72) | 93.50 (12.40) | 96.27 (7.62)

ADVERSE EVENTS:
Arm/Group | Remifentanil RS1 | Remifentanil RS2 | Meperidine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 7/30 | 9/30 | 16/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3.33% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remifentanil RS1 (N=30) | Remifentanil RS2 (N=30) | Meperidine (N=30)
Hypotension (Vascular disorders) | 5 | 4 | 6
Bradycardia (Cardiac disorders) | 2 | 1 | 1
Desaturation (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Dizziness (Ear and labyrinth disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Disinhibition (Psychiatric disorders) | 0 | 0 | 4
Amnesia (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No